CLINICAL TRIAL: NCT00105807
Title: The Effect of Exercise on Muscle, Function and Cost in VA Nursing Home Residents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: NRI 99-344
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: participation in low intensity exercise; Behavioral: participation in art and music activities

INTERVENTIONS:
Behavioral: participation in low intensity exercise
Behavioral: participation in art and music activities

SUMMARY:
Veterans are admitted to Veterans Health Administration (VA) Nursing Homes (NH) because impairment in their ability to perform activities of daily living (ADL) overwhelms their support system (family/friends) in the community. The etiologies of this impairment are, in part, due to chronic disease, deconditioning, and immobility. Yet, after admission, NH residents frequently have decreased levels of daily activity compared with their preadmission activity. Our preliminary observations suggest that dependent, frail residents improve in function in response to exercise in a NH setting.

DETAILED DESCRIPTION:
Background:

Veterans are admitted to Veterans Health Administration (VA) Nursing Homes (NH) because impairment in their ability to perform activities of daily living (ADL) overwhelms their support system (family/friends) in the community. The etiologies of this impairment are, in part, due to chronic disease, deconditioning, and immobility. Yet, after admission, NH residents frequently have decreased levels of daily activity compared with their preadmission activity. Our preliminary observations suggest that dependent, frail residents improve in function in response to exercise in a NH setting.

Objectives:

By comparing an exercise group with a non-exercise group that receives a comparable level of staff attention and positive reinforcement, we will determine whether changes in function normally associated with low intensity exercise are due to exercise or to other factors.

Methods:

We conducted a blinded, prospective, randomized, controlled, clinical investigation at a VA nursing home, comparing the effect of four months of low intensity exercise with the effect of music and art activity on: 1) muscle mass, assessed by DEXA scan; 2) physical function, assessed by timed performance tests, strength and independence in ADL; and 3) the cost of NH care, assessed by measuring the cost of providing care within the NH minus the cost of providing the intervention. Study setting is a VA nursing home, resident participants are new admissions to the NH and are 65 years or older. All participants must be able to follow a one step command and be able to participate in group activity. Participants with a Mini Mental Status Exam (MMSE) of less than 24/30 must have consent of authorized representative. Screening of candidates is completed on all NH admissions. Upon completion of the consent process, participants are randomly assigned to either the exercise group or the music/art group. Baseline tests including the DEXA scan, timed performance tests and observation of ADL is completed prior to participation in activity. At the conclusion of four months of activity, all baseline tests are repeated.

Status:

Recruitment and intervention stage of this project has been completed. In order to achieve our desired number of participants, a request was made and approval received for an extension of recruitment stage from March 2005 until December 2005. Interventions would continue through March 2006 and analysis of data completed in December 2006.

ELIGIBILITY:
Inclusion Criteria:

must be able to follow a one step command and be able to participate in group activity Participants with a Mini Mental Status Exam (MMSE) of less than 24/30 must have consent of authorized representative. Nursing Home resident

Exclusion Criteria:

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2002-07; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary M. Grant, BSN MA, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States